CLINICAL TRIAL: NCT04886076
Title: Circadian Rhythms Regulation in Pre-Manifest Synucleinopathies
Brief Title: Sleep Profiles in REM Sleep Behavior Disorder
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aleksandar Videnovic, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2018P000894
Record Dates: First submitted 2019-08-12; First posted 2021-05-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Rapid Eye Movement Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with RBD: Participants with REM Sleep Behavior Disorder
- Participants without RBD: Age- and gender-matched controls, without REM Sleep Behavior Disorder

SUMMARY:
Rapid eye movement (REM) sleep behavior disorder (RBD) is a sleep disorder in which you act out dreams during REM sleep. Sleep disturbances are very common in RBD, where they negatively impact patients' quality of life and safety. One of the known causes of sleep disturbance is the impairment of the "circadian rhythm", or the human sleep/wake cycle. The purpose of this study is to examine the role of disruption of the circadian rhythm in the development of RBD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RBD as assessed by the International Classification of Sleep Disorders (ICDS) diagnostic criteria within 3 years
2. 40 yrs of age

Exclusion Criteria:

1. Other significant neurological disorder
2. Untreated significant sleep apnea and/or current sleep apnea symptoms as assessed by the clinical investigator
3. Co-existent restless legs syndrome (RLS), as assessed by the ICDS diagnostic criteria for RLS
4. Cognitive impairment as determined by the Montreal Cognitive Assessment (MoCA) score of ≤ 23
5. Presence of depression defined as the Beck Depression Inventory (BDI) score >20
6. Use of tricyclic antidepressants, MAO inhibitors or selective serotonin reuptake inhibitors since they may induce/worsen RBD, unless on a stable dose of medication for at least 8 weeks
7. Use of medications known to affect melatonin secretion, such as lithium, α- and β-adrenergic antagonists
8. Shift work, currently or within the prior 3 months
9. Travel through ≥ 2 time zones within 60 days prior to the screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve men and women of all ethnic groups. We will recruit adults ≥ 40 years of age.
  Control participants will be age- (±5 years) and gender-matched to participants with RBD, have no diagnosis of RBD, and meet all other inclusion/inclusion criteria as the RBD group.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Circadian Amplitude | Study Day 17-18
  amplitude and area under the curve (AUC) of serum melatonin and clock gene expression
REM Sleep Phenomena | Study Day 16-17
  REM (rapid eye movement) sleep duration, REM Index, and EMG (electromyographic) activity) assessed via overnight Polysomnography
Objective Daytime Sleepiness | Study Day 17
  MSLT (Multiple Sleep Latency Test) assessed via Polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No